CLINICAL TRIAL: NCT03069547
Title: Comparative Effectiveness of Therapeutic Hip and Knee Exercise for Atellofemoral Pain: A Pragmatic Randomised Trial
Brief Title: Comparison of Exercise Therapies for Patellofemoral Pain
Acronym: COMPETE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FYS-2016-004
Record Dates: First submitted 2017-02-22; First posted 2017-03-03 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-08

CONDITIONS: Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Intervention Model Description: Eligible participants will be randomly assigned (1:1) to one of the two following groups:
  * QE - quadriceps exercise program
  * HE - hip exercise program
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators, study coordinators, outcome assessors, clinical staff, study staff, and other personnel directly involved in the clinical activities of the study, will be blinded to the group allocation.
  Participants and providers of the exercise delivery are not blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Quadriceps Exercise program (Active Comparator): The Quadricepts Exercise (QE) program runs for 12 weeks, with exercise sessions 3 times per week. Each training session is scheduled to last approximately 30 minutes. The exercise program is home based with monthly supervision visits at the clinic.
  Interventions: Other: Quadriceps Exercise program
- Hip Exercise program (Active Comparator): The Hip Exercise (HE) program runs for 12 weeks, with exercise sessions 3 times per week. Each training session is scheduled to last approximately 30 minutes. The exercise program is home based with monthly supervision visits at the clinic.
  Interventions: Other: Hip Exercise program

INTERVENTIONS:
Other: Quadriceps Exercise program — The exercise program is initiated at an individual clinical visit. An experienced physiotherapist introduces the participant to the exercise program and provides instructions to the individual exercises. An experienced physiotherapist provides the monthly supervision visits.
  The program details can be requested rom the responsible party. In brief the QE-program consists of:
  - A short warm-up and 3 specific exercises for the quadriceps muscle
  Progression of the exercise intensity is done by adding (additional) external loads, such as elastic rubber bands, free weights, etc.
  Arms: Quadriceps Exercise program
Other: Hip Exercise program — The exercise program is initiated at an individual clinical visit. An experienced physiotherapist introduces the participant to the exercise program and provides instructions to the individual exercises. An experienced physiotherapist provides the monthly supervision visits.
  The program details be requested rom the responsible party. In brief the HE-program consists of:
  - A short warm-up and 3 specific exercises for the hip abductor and extensor muscles
  Progression of the exercise intensity is done by adding (additional) external loads, such as elastic rubber bands, body weight etc.
  Arms: Hip Exercise program

SUMMARY:
Patellofemoral Pain (PFP) is a common knee problem, primarily affecting adolescents and young adults. PFP is characterised by significant retropatellar and/or peripatellar pain and impairment of function and quality of daily life. Exercise therapy is unequivocally recommended as a core component of the management of PFP. Different exercise types (e.g. quadriceps strengthening, hip strengthening and functional/neuromuscular exercises) have been investigated, with knee and hip strengthening exercises as the most common and recommended types. These exercises approaches produce similar small to moderate effects on pain and physical function. However, the PFP population is very heterogeneous and "one-size-fits-all"-approaches presumably are sub-optimal because the heterogeneity is ignored. The heterogeneity probably explains the overall limited beneficial effects of exercise, and the lack of differences in direct comparisons of different exercise types. In that sense, it is not unlikely that certain patient characteristics may predict outcome success of either a hip training program or a training program that focus on the quadriceps but this remains to be shown.

This study has two aims:

1. To assess the comparative effectiveness of two different exercise programs (Quadricep Exercise [QE] vs. Hip Exercise [HE]) on self-reported pain and function in individuals with PFP.
2. To explore candidate patient characteristics that predict differential responses to the two exercise programs (QE vs HE) on self-reported pain and physical function in individuals with PFP.

According to the study aims we pursue the following hypothesis:

- QE and HE have equivalent efficacy on self-reported pain after 12 weeks of treatment in patients with PFP.

The second study aim is to explore possible candidate patient characteristics that may associate with differential outcomes. As this is exploratory, the pursuit of this aim is hypothesis-free.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of PFP in at least one knee
* Visual analogue score rating of pain during activities of daily living during the previous week at a minimum of 3 on a 10 cm scale.
* Insidious onset of symptoms unrelated to trauma and persistent for at least 4 weeks.
* Pain in the anterior knee associated with at least 3 of the following:

  * During or after activity
  * Prolonged sitting
  * Stair ascent or descent
  * Squatting

Exclusion Criteria:

* Meniscal or other intra-articular injury
* Cruciate or collateral ligament laxity or tenderness
* Patellar tendon, iliotibial band, or pes anserine tenderness
* Osgood-Schlatter or Sinding-Larsen-Johansson syndrome
* History of recurrent patellar subluxation or dislocation
* History of surgery to the knee joint
* History of head injury or vestibular disorder within the last 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-04-10 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the KUJALA scoring questionnaire | week 12 and 26
  The Kujala Patellofemoral Scale - sometimes called the anterior knee pain scale - is disease specific validated disability scale ranging from 0 (complete disability) to 100 (fully functional). It is a 13-item self-report questionnaire that documents response to 6 activities (walking, running, jumping, climbing stairs, squatting, and sitting for prolonged periods with knees bent), as well as symptoms such as limp, inability to weight bear, swelling, abnormal patellar movement, muscle atrophy, and limitations in knee flexion.

SECONDARY OUTCOMES:
Change from baseline in the KOOS questionnaire | Week 12 and 26
  The Knee injury and Osteoarthritis Outcome Score (KOOS) is used to assess patient-reported knee-related symptoms. The KOOS is a patient-reported outcome measurement instrument developed to assess the patient's opinion about their knee and associated problems.KOOS comprises of 42 items in 5 separately scored subdomains: KOOS Pain (9 items), KOOS Symptoms (7 items), Function in daily living (KOOS Function; 17 items), Function in Sport and Recreation (5 items), and Knee-related Quality of Life (4 items). The previous week is the time period considered when answering the questions, and the questions relate to one knee (the target knee in this trial).
Change fom baseline in isometric muscle strength of hip abductors, hip external rotators, hip extensors, and quadriceps | Week 12
  Isometric muscle strength of hip abductors, hip external rotators, quadriceps, and hamstrings is performed by using a handheld dynamometer following a previously published testing protocol.
Change fom baseline in the Dynamic Assessment of Pain test | Week 12
  The Dynamic Assessment of Pain Test is a simple performance test with an integrated pain score, designed to provide useful information for monitoring treatment progress and evaluating treatment effects in clinical physiotherapy practice. The patient is asked to perform as many squatting movements (both legs) as possible within 30 seconds. The knees should reach approximately 90 degrees of flexion and full extension for each squat. This is supervised by the rater. There outcome of the test is the knee pain during the test on a 0-10 Numeric Rating Scale (NRS) rated immediately after the test.
Change fom baseline in the Pain Self-Efficacy Questionnaire | Week 12 and 26
  The pain self-efficacy questionnaire is a 10-item questionnaire developed to assess the confidence people with pain have in performing activities while in pain. It is applicable to all persisting pain presentations, and covers a range of functions. Confidence in performing activities are rated on a 7-point (0-6) Likert scale with 0 representing not at all confident and 6 representing completely confident. A total score is calculated by summing the answers producing a score between 0 and 60. Higher scores reflect stronger self-efficacy beliefs.
Change fom baseline in the EuroQoL Questionnaire | Week 12 and 26
  The EuroQoL questionnaire is a standardised patient-reported instrument for use as a measure of health related quality of life.
Transition Questionnaire of global perceived effect on overall health, pain, and function | Week 12 and 26
  The Transition Questionnaire of global perceived effect is an adaptive questionnaire in which the participants initially answer if their current state is "unchanged, worse" or "better" compared to the baseline visit. An "unchanged" equals a transition score of 0. If the participant answers "worse", he/she is asked to rate the degree of worsening on a 7 point Likert scale, and the corresponding scores range from -1 to -7. Correspondingly, if a participant answers "better", he/she is asked to rate the degree of improvement on a 7 point Likert scale, and the corresponding scores range from 1 to 7. Thus the Transition score range from -7 (worsening) to 7 (improvement), with the mid-point - 0 - representing no change. The transition scale is used to assess overall knee related health status.

OTHER OUTCOMES:
Candidate prognostic factor: Previous treatments received | Baseline (week 0)
  Participants are surveyed about any previous treatments they have received for their current PFP (target knee only)
Candidate prognostic factor: Presence of bilateral knee pain | Baseline (week 0)
  Self-reported presence and frequency of pain in the contralateral knee (not target knee). The participants are asked to estimate the frequency of pain in contralateral knee pain during that last 3 months. Predefined frequency options are available:
  * Almost daily
  * Several times during a week
  * Weekly
  * Monthly
  * Rarely
  We will a priori define a dichotomisation of the scores as "frequent bilateral knee pain" ("Almost daily" and "several times during a week") and "infrequent bilateral knee pain" ("Weekly", "Monthly", and "Rarely"). We will make sensitivity tests of this a priori cut-off by changing the cut-off value by +/- frequency option.
Candidate prognostic factor: Presence of pain in other lower extremity joints (feet, ankles, hips) | Baseline (week 0)
  Self-reported presence of pain in the feet, ankles, and/or hips lasting more than 3 months, recorded as "Yes" (pain present) or "No" (No pain) for feet, ankles and hips, respectively. The participants are asked to estimate the frequency of pain in other lower extremity joints (feet, ankles, and hips) during that last 3 months. Predefined frequency options are available:
  * Almost daily
  * Several times during a week
  * Weekly
  * Monthly
  * Rarely
  We will a priori define a dichotomisation of the scores as "frequent [foot/ankle/hip] pain" ("Almost daily" and "several times during a week") and "infrequent [foot/ankle/hip] pain" ("Weekly", "Monthly", and "Rarely"). We will make sensitivity tests of this a priori cut-off by changing the cut-off value by +/- frequency option.
Candidate prognostic factor: Presence of low back pain | Baseline (week 0)
  Self-reported presence and frequency of low back pain. The participants are asked to estimate the frequency of low back pain during that last 3 months. Predefined frequency options are available:
  * Almost daily
  * Several times during a week
  * Weekly
  * Monthly
  * Rarely
  We will a priori define a dichotomisation of the scores as "frequent low back pain" ("Almost daily" and "several times during a week") and "infrequent low back pain" ("Weekly", "Monthly", and "Rarely"). We will make sensitivity tests of this a priori cut-off by changing the cut-off value by +/- frequency option.
Candidate prognostic factor: PainDetect questionnaire | Baseline (week 0)
  The painDETECT questionnaire (PDQ) is a patient reported questionnaire developed and validated to assess presence of signs of neuropathic pain. It comprises questions regarding pain intensity, course of pain, subjective experience of a radiating quality of the pain, and the presence and perceived severity of seven somatosensory symptoms of neuropathic pain. A validated algorithm is used to calculate a total score ranging from 0 to 38. A score ≤12 indicates that the presence of neuropathic pain is unlikely, a score ≥19 indicates that a neuropathic pain component is likely to be present, while a score of 13-18 points towards unclear screening conclusion.
Candidate prognostic factor: Exercise Self-Efficacy Questionnaire | Baseline (week 0)
  Exercise self-efficacy in relation to the two different exercise programs are assessed by asking the participants to rate their confidence in performing the two different exercise programs on a 7-point (0-6) Likert scale with 0 representing "Not at all confident" and 6 representing "Completely confident".
Candidate prognostic factor: Pain Catastrophizing Scale | Baseline (week 0)
  The Pain Catastrophizing Scale (PCS) will used as a measure of pain-related catastrophic thinking. The PCS instructs participants to reflect upon past painful experiences, and to indicate the frequency with which 13 pre-specified thoughts or feelings occur while they are experiencing pain. The frequency is scored on a 5-point scale ranging from 0 (not at all) to 4 (all the time). The PCS measures 3 distinct components: rumination, magnification, and helplessness.
Candidate prognostic factor: Hyper mobility | Baseline (week 0)
  Hypermobility is assessed by the Beighton Score (28) applying the revised criteria for the diagnosis of benign joint hypermobility syndrome. The Beighton score ranges from 0-9. In this study we define hypermobility as a score of 4 or more.
Candidate prognostic factor: Knee joint alignment during a forward lunge | Baseline (week 0)
  Knee joint alignment is assessed by clinically observation of the participant while he/she performs a forward lunge movement. The observation is made by a trained physiotherapist that classifies each participant's knee as "varus", "neutral", or "valgus".
Candidate prognostic factor: Knee joint alignment during a single-leg mini-squat | Baseline (week 0)
  Knee joint alignment is assessed by clinically observation of the participant while he/she performs a single-leg mini-squat movement. The observation is made by a trained physiotherapist that classifies each participant's knee as "varus", "neutral", or "valgus".
Candidate prognostic factor: Physiotherapist assessed prognosis for the participant based on group allocation | Baseline (week 0)
  A trained physiotherapist's estimate of each patient's potential for a successful outcome based on professional appraisal. The therapists are instructed to score each patient on a continuum of 1 (suggesting a very poor projected outcome) to 10 (suggesting an excellent projected outcome). The therapist must score each patient following their complete encounter with the patient. This may include the physiotherapist's assessment of the patient's resources (personal, material, social, etc.), personality, medical history, comorbidities, surgery reports, physical examination(s), physiotherapeutic assessments, and more.
Candidate prognostic factor: Midfoot mobility | Baseline (week 0)
  Midfoot mobility is calculated as the change in midfoot width from non-weight bearing to weight bearing. Midfoot width is measured at 50% of total foot length using a caliper during non-weight bearing and during standing with equal weight on each foot. The mobility is recorded as the difference between non-weight bearing and weight bearing measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Marius Henriksen, PT, PhD, Study Chair — Department of Physical and Occupational Therapy, Bispebjerg-Frederiksberg Hospital
Locations (1):
- Bispebjerg Hospital, Department of Physical and Occupational Therapy, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared once the study is finalised and results pulished. IPD can be obtained by contacting the responsible party

REFERENCES:
- [Derived] Hansen R, Rathleff MS, Brushoj C, Magnusson SP, Henriksen M. Differential Effects of Quadriceps and Hip Muscle Exercises for Patellofemoral Pain: A Secondary Effect Modifier Analysis of a Randomized Trial. J Orthop Sports Phys Ther. 2024 Nov;54(11):732-742. doi: 10.2519/jospt.2024.12503. PMID 39478429
- [Derived] Jorgensen JEV, Rathleff MS, Henriksen M, Brushoj C, Hansen R. Physical Therapists' Prognosis of Outcomes After a Hip or Quadriceps Exercise Intervention in Patients With Patellofemoral Pain: A Secondary Analysis of a Randomized Trial. J Orthop Sports Phys Ther. 2024 Aug;54(8):541-550. doi: 10.2519/jospt.2024.12258. PMID 38840581
- [Derived] Hansen R, Brushoj C, Rathleff MS, Magnusson SP, Henriksen M. Quadriceps or hip exercises for patellofemoral pain? A randomised controlled equivalence trial. Br J Sports Med. 2023 Oct;57(20):1287-1294. doi: 10.1136/bjsports-2022-106197. Epub 2023 May 3. PMID 37137673

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-10-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT03069547/SAP_000.pdf